CLINICAL TRIAL: NCT03992638
Title: Mechanisms of LPRF Action in the Promotion of Wound Healing and Tissue Regeneration: A Randomised Controlled Trial
Brief Title: Mechanisms of LPRF Action in the Promotion of Wound Healing and Tissue Regeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The European Research Group on Periodontology (ERGOPerio) (Network)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Maurizio Tonetti, Executive Director, Clinical Professor, The European Research Group on Periodontology (ERGOPerio)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Perio20190614
Record Dates: First submitted 2019-06-17; First posted 2019-06-20 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Leukocyte Count

STUDY DESIGN:
Intervention Model Description: Split-mouth design allowing to assess two types of treatment in the same patient.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-PRF membrane (Experimental): Periodontal plastic surgical procedures (coronally advanced flap, CAF) in combination with a double layer autologous leucocyte and platelet-rich fibrin (L-PRF) membrane.
  Interventions: Procedure: leucocyte and platelet-rich fibrin (L-PRF) in combination with CAF
- Control (Active Comparator): CAF
  Interventions: Procedure: CAF

INTERVENTIONS:
Procedure: leucocyte and platelet-rich fibrin (L-PRF) in combination with CAF — Completing root coverage by coronally advanced flap technique in combination with L-PRF.
  Arms: L-PRF membrane
Procedure: CAF — Completing root coverage by coronally advanced flap technique alone
  Arms: Control

SUMMARY:
This study evaluates the clinical and biological effects of leucocyte and platelet-rich fibrin (L-PRF) on intraoral wound healing.

DETAILED DESCRIPTION:
Gingival recession is characterized by the exposure of root surfaces of the tooth, is attributed to the apical migration of the gingival marginal tissue, and it is a frequently noted clinical feature in all populations. Other than cosmetic problems, a gingival recession can have a causative role in tooth sensitivity, and contribute to difficulties in oral hygiene maintenance or root caries. Moreover, it may worsen with time.

The ultimate goal of surgical root-coverage procedures (Periodontal plastic surgery) is the elimination of the recession defect with minimal probing depths after treatment, along with the ability to restore the natural color and texture of the gingiva (gum). By achieving root coverage, overall improved aesthetics, prevention of non-carious cervical lesions or root caries, and treatment of the resulting root sensitivity should be expected.

Surgical interventions in general, and in particular those aiming to reconstruct tissues lost due to trauma or disease in particular, are biologically dependent on a cascade of unimpaired wound healing mechanisms, including a non-disrupted inflammatory process, vascularization(blood supply) of the wound area, and consequent tissue regeneration. Wound healing has been defined as "the natural response to injury compiling a cascade of complex events orchestrated in a way that many cell types guided by the release of soluble mediators and signals. In a bid to enhance this phase, autologous platelet 'concentrates' were developed, derived from centrifuged blood of patients and applied as surgical adjuncts. Previous studies indicate that leucocyte plasma rich fibrin (LPRF/newest generation of platelet concentrates) preparations significantly modulate wound healing and promote tissue regeneration in a variety of oral surgical procedures. Clinical studies where LPRF is analyzed at the molecular level to quantify the temporal release of growth factors, cytokines, or other biomolecular components are still lacking. Despite the broad application of LPRF in modern dentistry information which integrates clinical and molecular data from in vivo models are essential to elucidate its relevant biological mechanisms. The mechanisms of action are unclear, and the relative role of their different components have not been fully explained. This study will aim to investigate if LPRF can offer superior clinical outcomes and will compare the concentrations and kinetics of wound healing regulators in root coverage procedures with and without local application of LPRF.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Non-smokers or former smokers
* Participants must agree to read the "Patient information leaflet and provide a signed a copy of the "Informed Consent", after the study design has been completely explained.
* Presence of bilateral isolated Miller Class I and II gingival recessions in anterior and premolar regions.
* Presence of minimum 2 mm of keratinized gingiva apical to the gingival margin at the selected sites.

Exclusion Criteria:

* The patient is medically compromised with history of diabetes mellitus or hepatic or renal disease, or other serious medical conditions or transmittable diseases e.g. Hepatitis B or C or AIDS.
* History of rheumatic fever, heart murmur, mitral valve prolapse, artificial heart valve or conditions which would require antibiotic prophylaxis invasive dental procedures.
* Patients undergoing therapies involving the use of antibiotic, anti-inflammatory or anticoagulant drugs during the month prior to the baseline exam.
* History of alcohol use or drug abuse.
* Self-reported pregnancy or lactation.
* Subjects would be considered inappropriate for the trial if they have a history of pre-existing acute or chronic medical or psychiatric illness and laboratory abnormality which may pose to increase the risk of the subjects involved in the trial or administering the investigational product or may interfere with the interpretation of trial results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change of gingival recession depth (GR) from baseline to 6 months | Baseline, 3 months, and 6 months
  Measured from the CEJ to the apical extension of the gingival margin in mm with the use of Florida probe.
Change of probing pocket depth (PPD) from baseline to 6 months | Baseline, 3 months, and 6 months
  Measured from the gingival margin to base of the gingival sulcus in mm with the use of Florida probe.
Change of clinical attachment level (CAL) from baseline to 6 months | Baseline, 3 months, and 6 months
  Measured from cementoenamel junction (CEJ) to the base of the gingival sulcus in mm with the use of Florida probe.
Change of keratinized mucosa width (KMW) from baseline to 6 months | Baseline, 3 months, and 6 months
  Measured from the gingival margin to the mucogingival line in mm with the use of Florida probe.
Change of thickness of keratinised gingiva (GT) from baseline to 6 months | Baseline, 3 months, and 6 months
  Measured 3 mm apical to the gingival margin in mm measured by superimposition of intraoral digital scanning images.

SECONDARY OUTCOMES:
Concentration of gingival wound fluid molecules | Baseline, 6 hours, 3 days, and 7 days
  Concentration changes of the molecules and inflammatory mediators in the wound fluid (WF).

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Tonetti, PhD MMSc, Principal Investigator — The European Research Group on Periodontology (ERGOPerio)
Locations (1):
- Faculty of Dentistry, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agudio G, Nieri M, Rotundo R, Franceschi D, Cortellini P, Pini Prato GP. Periodontal conditions of sites treated with gingival-augmentation surgery compared to untreated contralateral homologous sites: a 10- to 27-year long-term study. J Periodontol. 2009 Sep;80(9):1399-405. doi: 10.1902/jop.2009.090122. PMID 19722789
- [Background] Aroca S, Keglevich T, Barbieri B, Gera I, Etienne D. Clinical evaluation of a modified coronally advanced flap alone or in combination with a platelet-rich fibrin membrane for the treatment of adjacent multiple gingival recessions: a 6-month study. J Periodontol. 2009 Feb;80(2):244-52. doi: 10.1902/jop.2009.080253. PMID 19186964
- [Background] Cairo F, Pagliaro U, Nieri M. Treatment of gingival recession with coronally advanced flap procedures: a systematic review. J Clin Periodontol. 2008 Sep;35(8 Suppl):136-62. doi: 10.1111/j.1600-051X.2008.01267.x. PMID 18724847
- [Background] Cairo F, Rotundo R, Miller PD, Pini Prato GP. Root coverage esthetic score: a system to evaluate the esthetic outcome of the treatment of gingival recession through evaluation of clinical cases. J Periodontol. 2009 Apr;80(4):705-10. doi: 10.1902/jop.2009.080565. PMID 19335093
- [Background] Cardaropoli D, Tamagnone L, Roffredo A, Gaveglio L. Treatment of gingival recession defects using coronally advanced flap with a porcine collagen matrix compared to coronally advanced flap with connective tissue graft: a randomized controlled clinical trial. J Periodontol. 2012 Mar;83(3):321-8. doi: 10.1902/jop.2011.110215. Epub 2011 Jul 1. PMID 21721988
- [Background] Castro AB, Meschi N, Temmerman A, Pinto N, Lambrechts P, Teughels W, Quirynen M. Regenerative potential of leucocyte- and platelet-rich fibrin. Part A: intra-bony defects, furcation defects and periodontal plastic surgery. A systematic review and meta-analysis. J Clin Periodontol. 2017 Jan;44(1):67-82. doi: 10.1111/jcpe.12643. Epub 2016 Nov 24. PMID 27783851
- [Background] Chambrone L, Lima LA, Pustiglioni FE, Chambrone LA. Systematic review of periodontal plastic surgery in the treatment of multiple recession-type defects. J Can Dent Assoc. 2009 Apr;75(3):203a-203f. PMID 19356319
- [Background] Clauser C, Nieri M, Franceschi D, Pagliaro U, Pini-Prato G. Evidence-based mucogingival therapy. Part 2: Ordinary and individual patient data meta-analyses of surgical treatment of recession using complete root coverage as the outcome variable. J Periodontol. 2003 May;74(5):741-56. doi: 10.1902/jop.2003.74.5.741. PMID 12816306
- [Background] Clipet F, Tricot S, Alno N, Massot M, Solhi H, Cathelineau G, Perez F, De Mello G, Pellen-Mussi P. In vitro effects of Choukroun's platelet-rich fibrin conditioned medium on 3 different cell lines implicated in dental implantology. Implant Dent. 2012 Feb;21(1):51-6. doi: 10.1097/ID.0b013e31822b9cb4. PMID 21986450
- [Background] Cortellini P, Pini Prato G. Coronally advanced flap and combination therapy for root coverage. Clinical strategies based on scientific evidence and clinical experience. Periodontol 2000. 2012 Jun;59(1):158-84. doi: 10.1111/j.1600-0757.2011.00434.x. PMID 22507065
- [Background] Culhaoglu R, Taner L, Guler B. Evaluation of the effect of dose-dependent platelet-rich fibrin membrane on treatment of gingival recession: a randomized, controlled clinical trial. J Appl Oral Sci. 2018 May 14;26:e20170278. doi: 10.1590/1678-7757-2017-0278. PMID 29768524
- [Background] Dohan Ehrenfest DM, Andia I, Zumstein MA, Zhang CQ, Pinto NR, Bielecki T. Classification of platelet concentrates (Platelet-Rich Plasma-PRP, Platelet-Rich Fibrin-PRF) for topical and infiltrative use in orthopedic and sports medicine: current consensus, clinical implications and perspectives. Muscles Ligaments Tendons J. 2014 May 8;4(1):3-9. eCollection 2014 Jan. PMID 24932440
- [Background] Del Pizzo M, Zucchelli G, Modica F, Villa R, Debernardi C. Coronally advanced flap with or without enamel matrix derivative for root coverage: a 2-year study. J Clin Periodontol. 2005 Nov;32(11):1181-7. doi: 10.1111/j.1600-051X.2005.00831.x. PMID 16212581
- [Background] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part I: technological concepts and evolution. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e37-44. doi: 10.1016/j.tripleo.2005.07.008. Epub 2006 Jan 19. PMID 16504849
- [Background] Dos Santos Canellas JV, Ritto FG, Medeiros PJD. Efficacy of Platelet-Rich Fibrin After Mandibular Third Molar Extraction: A Systematic Review and Meta-Analysis. J Oral Maxillofac Surg. 2017 Aug;75(8):1576-1577. doi: 10.1016/j.joms.2017.03.060. Epub 2017 May 15. No abstract available. PMID 28521145
- [Background] Giannobile WV, Lynch SE, Denmark RG, Paquette DW, Fiorellini JP, Williams RC. Crevicular fluid osteocalcin and pyridinoline cross-linked carboxyterminal telopeptide of type I collagen (ICTP) as markers of rapid bone turnover in periodontitis. A pilot study in beagle dogs. J Clin Periodontol. 1995 Dec;22(12):903-10. doi: 10.1111/j.1600-051x.1995.tb01793.x. PMID 8613557
- [Background] Guo S, Dipietro LA. Factors affecting wound healing. J Dent Res. 2010 Mar;89(3):219-29. doi: 10.1177/0022034509359125. Epub 2010 Feb 5. PMID 20139336
- [Background] Kassab MM, Cohen RE. The etiology and prevalence of gingival recession. J Am Dent Assoc. 2003 Feb;134(2):220-5. doi: 10.14219/jada.archive.2003.0137. PMID 12636127
- [Background] Kobayashi E, Fluckiger L, Fujioka-Kobayashi M, Sawada K, Sculean A, Schaller B, Miron RJ. Comparative release of growth factors from PRP, PRF, and advanced-PRF. Clin Oral Investig. 2016 Dec;20(9):2353-2360. doi: 10.1007/s00784-016-1719-1. Epub 2016 Jan 25. PMID 26809431
- [Background] Liu F, Pelekos G, Jin LJ. The gingival biotype in a cohort of Chinese subjects with and without history of periodontal disease. J Periodontal Res. 2017 Dec;52(6):1004-1010. doi: 10.1111/jre.12471. Epub 2017 Jun 15. PMID 28617953
- [Background] Loe H, Anerud A, Boysen H. The natural history of periodontal disease in man: prevalence, severity, and extent of gingival recession. J Periodontol. 1992 Jun;63(6):489-95. doi: 10.1902/jop.1992.63.6.489. PMID 1625148
- [Background] de Sanctis M, Zucchelli G. Coronally advanced flap: a modified surgical approach for isolated recession-type defects: three-year results. J Clin Periodontol. 2007 Mar;34(3):262-8. doi: 10.1111/j.1600-051X.2006.01039.x. PMID 17309597
- [Background] Marx RE, Carlson ER, Eichstaedt RM, Schimmele SR, Strauss JE, Georgeff KR. Platelet-rich plasma: Growth factor enhancement for bone grafts. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1998 Jun;85(6):638-46. doi: 10.1016/s1079-2104(98)90029-4. PMID 9638695
- [Background] Masuki H, Okudera T, Watanebe T, Suzuki M, Nishiyama K, Okudera H, Nakata K, Uematsu K, Su CY, Kawase T. Growth factor and pro-inflammatory cytokine contents in platelet-rich plasma (PRP), plasma rich in growth factors (PRGF), advanced platelet-rich fibrin (A-PRF), and concentrated growth factors (CGF). Int J Implant Dent. 2016 Dec;2(1):19. doi: 10.1186/s40729-016-0052-4. Epub 2016 Aug 22. PMID 27747711
- [Background] Moraschini V, Barboza Edos S. Use of Platelet-Rich Fibrin Membrane in the Treatment of Gingival Recession: A Systematic Review and Meta-Analysis. J Periodontol. 2016 Mar;87(3):281-90. doi: 10.1902/jop.2015.150420. Epub 2015 Nov 12. PMID 26561997
- [Background] Naik B, Karunakar P, Jayadev M, Marshal VR. Role of Platelet rich fibrin in wound healing: A critical review. J Conserv Dent. 2013 Jul;16(4):284-93. doi: 10.4103/0972-0707.114344. PMID 23956527
- [Background] Pellegrini G, Rasperini G, Pagni G, Giannobile WV, Milani S, Musto F, Dellavia C. Local wound healing biomarkers for real-time assessment of periodontal regeneration: pilot study. J Periodontal Res. 2017 Jun;52(3):388-396. doi: 10.1111/jre.12403. Epub 2016 Aug 11. PMID 27510312
- [Background] Pini Prato GP, Baldi C, Nieri M, Franseschi D, Cortellini P, Clauser C, Rotundo R, Muzzi L. Coronally advanced flap: the post-surgical position of the gingival margin is an important factor for achieving complete root coverage. J Periodontol. 2005 May;76(5):713-22. doi: 10.1902/jop.2005.76.5.713. PMID 15898931
- [Background] Miron RJ, Zucchelli G, Pikos MA, Salama M, Lee S, Guillemette V, Fujioka-Kobayashi M, Bishara M, Zhang Y, Wang HL, Chandad F, Nacopoulos C, Simonpieri A, Aalam AA, Felice P, Sammartino G, Ghanaati S, Hernandez MA, Choukroun J. Use of platelet-rich fibrin in regenerative dentistry: a systematic review. Clin Oral Investig. 2017 Jul;21(6):1913-1927. doi: 10.1007/s00784-017-2133-z. Epub 2017 May 27. PMID 28551729
- [Background] Roy S, Driggs J, Elgharably H, Biswas S, Findley M, Khanna S, Gnyawali U, Bergdall VK, Sen CK. Platelet-rich fibrin matrix improves wound angiogenesis via inducing endothelial cell proliferation. Wound Repair Regen. 2011 Nov;19(6):753-66. doi: 10.1111/j.1524-475X.2011.00740.x. PMID 22092846
- [Background] Serino G, Wennstrom JL, Lindhe J, Eneroth L. The prevalence and distribution of gingival recession in subjects with a high standard of oral hygiene. J Clin Periodontol. 1994 Jan;21(1):57-63. doi: 10.1111/j.1600-051x.1994.tb00278.x. PMID 8126246
- [Background] Temmerman A, Vandessel J, Castro A, Jacobs R, Teughels W, Pinto N, Quirynen M. The use of leucocyte and platelet-rich fibrin in socket management and ridge preservation: a split-mouth, randomized, controlled clinical trial. J Clin Periodontol. 2016 Nov;43(11):990-999. doi: 10.1111/jcpe.12612. Epub 2016 Sep 21. PMID 27509214
- [Background] Zucchelli G, Mounssif I. Periodontal plastic surgery. Periodontol 2000. 2015 Jun;68(1):333-68. doi: 10.1111/prd.12059. PMID 25867992